CLINICAL TRIAL: NCT05254288
Title: Evaluation of a New In-office and Domiciliary Ozonized Gel for the Management of Periodontal Disease
Brief Title: In-office and Domiciliary Use of a New Ozonized Gel for the Management of Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-OZORALPAROD
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Periodontal Diseases
Keywords: ozone; chlorhexidine; split-mouth
MeSH Terms: conditions — Periodontal Diseases | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Split-mouth
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Gels concealed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split-mouth Group A (Experimental): Half of patients will be assigned to this group. Quadrants Q1/Q4 will receive ozone administration. Quadrants Q2/Q3 will receive chlorhexidine administration.
  Interventions: Other: Chlorhexidine; Other: Ozoral gels
- Split-mouth Group B (Experimental): Half of patients will be assigned to this group Quadrants Q2/Q3 will receive ozone administration. Quadrants Q1/Q4 will receive chlorhexidine administration.
  Interventions: Other: Chlorhexidine; Other: Ozoral gels

INTERVENTIONS:
Other: Chlorhexidine — In-office and domiciliary use of chlorhexidine for 14 days.
Other: Ozoral gels — In-office administration of Ozoral Pro and domiciliary use of Ozoral gel for 14 days.

SUMMARY:
The aim of this study is to evaluate the efficacy of non-surgical periodontal therapy with supportive home oral care for the treatment of periodontal disease.

Patients with bilateral periodontal pathological sites will undergo professional dental hygiene with ultrasonic handpiece (Piezon EMS with PerioSlim inserts) followed by manual instrumentation with Gracey curettes and application of erythritol Airflow powders. Then, patients will be randomly divided into two groups according to a split-mouth design: the Control Group will undergo a split-mouth application of chlorhexidine gel 1% for quadrants 1/3 (or 2/4), while for the Trial Group Ozoral Pro for quadrants 2/4 (or 1/3) will be used. Patients will use the products at home with one daily application for the following 14 days after the visits. The Trial Group will use Ozoral Gel for home applications.

The following indexes will be assessed at baseline, T1 (1 month), T2 (3 months) and T3 (6 months): recession, PPD, BoP %, CAL, PCR %. Contextually, the application of the two gels will be performed.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of non-surgical periodontal therapy with supportive home oral care for the treatment of periodontal disease comparing chlorhexidine and ozone gels.

Patients with bilateral periodontal pathological sites will undergo professional dental hygiene with ultrasonic handpiece (Piezon EMS with PerioSlim inserts) followed by manual instrumentation with Gracey curettes and application of erythritol Airflow powders. Then, patients will be randomly divided into two groups according to a split-mouth design:

* Control Group: application of chlorhexidine gel 1% for quadrants 1/3 (or 2/4)
* Trial Group: administration of Ozoral Pro for quadrants 2/4 (or 1/3).

Patients will use the products at home with one daily application for the following 14 days after the visits. The Trial Group will use Ozoral Gel for home applications.

The following indexes will be assessed at baseline, T1 (1 month), T2 (3 months) and T3 (6 months): recession, PPD, BoP %, CAL, PCR %. Contextually, the application of the two gels will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of bilateral periodontal sites according to the new Classification of Periodontal and Peri-implant Diseases (Severity: Staging I; Complexity: Staging II).
* No systemic disease;
* Compliant patients.

Exclusion Criteria:

* Absence of dental implants;
* Neurological and psychiatric diseases;
* Patients taking bisphosphonates during the previous 12 months from the beginning of the study;
* Pregnant and/or breastfeeding women;
* Patients undergoing anticancer therapy.
* Patients with poor compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Change in R - Gingival recession | Time Frame: baseline, 1, 3 and 6 months after baseline
  Distance (in mm) between the gingival margin and the amelo-cemental junction.
Change in PPD - Probing Pocket Depth | Time Frame: baseline, 1, 3 and 6 months after baseline
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in Bleeding on Probing (BOP%) | Time Frame: baseline, 1, 3 and 6 months after baseline
  Dichotomous scoring (yes/no) of bleeding sites
Change in Plaque Control Record (PCR%) | Time Frame: baseline, 1, 3 and 6 months after baseline
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.
Change in Dental mobility (Miller, 1985) | Time Frame: baseline, 1, 3 and 6 months after baseline
  Scoring criteria
  * Grade 0: oscillation within 0.2 mm; the teeth move naturally and there are no mobility problems;
  * Grade I: horizontal mobility of the tooth from 0.2 to 1 mm;
  * Grade II: horizontal mobility of the tooth from 1 to 2 mm;
  * Grado III: horizontal mobility equal to or greater than 3 mm or vertical mobility of the tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.